CLINICAL TRIAL: NCT01992874
Title: A Multi-Center, Open-Label, Single 60 mg Dose, Two Period, Two Sequence Cross-Over Trial to Investigate the Relative Bioavailability of Two Solid Oral Pimasertib Formulations in Cancer Patients
Brief Title: Relative Bioavailability of Pimasertib in Cancer Patients
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: EMD Serono (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Treatment
Other Study IDs: 200066-013
Record Dates: First submitted 2013-11-08; First posted 2013-11-25 (Estimated); Results first posted 2016-05-11 (Estimated); Last update posted 2017-08-15 (Actual); Status verified 2017-07

CONDITIONS: Neoplasms
Keywords: Neoplasms; Pimasertib; Cancer
MeSH Terms: conditions — Neoplasms | interventions — N-(2,3-dihydroxypropyl)-1-((2-fluoro-4-iodophenyl)amino)isonicotinamide

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Pimasertib Capsule/Pimasertib Tablet (Experimental)
  Interventions: Drug: Pimasertib Capsule (Part A); Drug: Pimasertib Tablet (Part A); Drug: Pimasertib Capsule (Part B and trial extension phase)
- Pimasertib Tablet/Pimasertib Capsule (Experimental)
  Interventions: Drug: Pimasertib Tablet (Part A); Drug: Pimasertib Capsule (Part A); Drug: Pimasertib Capsule (Part B and trial extension phase)

INTERVENTIONS:
Drug: Pimasertib Capsule (Part A) — Pimasertib capsule administration at a single dose of 60 milligram (mg) orally on Day 1 in Part A.
  Other Names: AS703026; MSC1936369B
  Arms: Pimasertib Capsule/Pimasertib Tablet
Drug: Pimasertib Tablet (Part A) — Pimasertib tablet administration at a single dose of 60 mg orally on Day 3 in Part A.
  Other Names: AS703026; MSC1936369B
  Arms: Pimasertib Capsule/Pimasertib Tablet
Drug: Pimasertib Tablet (Part A) — Pimasertib tablet administration at a single dose of 60 mg orally on Day 1 in Part A.
  Other Names: AS703026; MSC1936369B
  Arms: Pimasertib Tablet/Pimasertib Capsule
Drug: Pimasertib Capsule (Part A) — Pimasertib capsule administration at a single dose of 60 mg orally on Day 3 in Part A.
  Other Names: AS703026; MSC1936369B
  Arms: Pimasertib Tablet/Pimasertib Capsule
Drug: Pimasertib Capsule (Part B and trial extension phase) — Subjects completing Part A to receive pimasertib capsule at a dose of 60 mg orally twice daily in cycles of 21 days each in Part B and trial extension phase until disease progression, intolerable toxicity, subject withdrawal, loss to follow-up or death.
  Other Names: AS703026; MSC1936369B

SUMMARY:
This is a Phase 1, multi-center, open-label, single-dose, 2 period, 2 sequence cross-over trial to investigate the relative bioavailability of 2 solid oral pimasertib formulations in cancer subjects (Part A), followed by open-label pimasertib administration (Part B and trial extension phase).

ELIGIBILITY:
Inclusion Criteria:

* Pathologically confirmed solid tumors, either refractory to standard therapy or for which no effective standard therapy is available, with a measurable disease as defined by Response Evaluation Criteria in Solid Tumors (RECIST) v1.1
* An Eastern Cooperative Oncology Group Performance Status (ECOG PS) of less than or equal to (<=) 1
* Other protocol defined inclusion criteria could apply

Exclusion Criteria:

* Disease conditions or concomitant medication that may significantly influence the conduct of the trial or an abnormal electrocardiogram (ECG) or blood pressure at Screening as defined in the protocol
* Treatment with strong inhibitors or inducers of cytochrome P450 2C19 (CYP2C19) and CYP3A4 including fruit juices or beverages containing these substances
* History of prior mitogen-activated protein kinase/extracellular signal-regulated kinase (MAPK/ERK) kinase (MEK) inhibitor exposure (including, pimasertib) or progression of disease on MEK inhibitors
* Evidence of a retinal vein occlusion (RVO) on fluorescein angiogram or a history of RVO
* Life expectancy of less than 12 weeks
* Other protocol defined exclusion criteria could apply

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 38 (Actual)
Dates: Start 2013-11-30 (Actual); Primary Completion 2014-05-31 (Actual); Study Completion 2015-02-28 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Medical Responsible, Study Director — EMD Serono, Inc., Rockland MA, a subsidiary of Merck KGaA, Darmstadt, Germany
Locations (1):
- Please Contact U.S. Medical Information Located in, Rockland, Massachusetts, United States

REFERENCES:
- [Result] Mahadevan D, Mita M, Richards D, McClay E, Heist RS, Kumar A, Sundararajan S, Naing A. Phase I single dose, two-period and two-sequence cross-over trial to evaluate the relative bioavailability of two oral pimasertib formulations in advanced cancer patients. Cancer Chemother Pharmacol. 2017 Apr;79(4):681-688. doi: 10.1007/s00280-017-3258-0. Epub 2017 Mar 13. PMID 28289865

RESULTS

PARTICIPANT FLOW:
Recruitment Details: First/last subject (informed consent): Nov 2013/Feb 2015. Clinical data cut-off: May 2014, Study completion date: Feb 2015
Pre-assignment Details: A total of 45 subjects were screened. 38 subjects were enrolled and received the trial medication completed two sequence cross-over Part A and further continued in open label Part B.
Groups:
- Part A: Pimasertib Capsule Then Pimasertib Tablet: A single dose of 2 Pimasertib 30 mg capsule administered orally on Day 1 in first intervention period followed by a single dose of 3 Pimasertib 20 mg tablet single dose administered orally on Day 3, of Part A of the study. A washout period of 48 hours was maintained between the administration of the two treatments.
- Part A: Pimasertib Tablet Then Pimasertib Capsule: A single dose of 3 Pimasertib 20 mg tablet administered orally on Day 1 in first intervention period followed by a single dose of 2 Pimasertib 30 mg capsule single dose administered orally on Day 3, of Part A of the study. A washout period of 48 hours was maintained between the administration of the two treatments.
- Part B:Pimasertib Capsule: Pimasertib 2 capsule 30 mg orally twice daily up to 4 cycles of 21 days each in Part B and trial extension phase until disease progression, intolerable toxicity, subject withdrawal, loss to follow-up or death.
Period: Part A
Arm/Group | Part A: Pimasertib Capsule Then Pimasertib Tablet | Part A: Pimasertib Tablet Then Pimasertib Capsule | Part B:Pimasertib Capsule
Started | 21 | 17 | 0
Completed | 21 | 17 | 0
Not Completed | 0 | 0 | 0
Period: Part B
Arm/Group | Part A: Pimasertib Capsule Then Pimasertib Tablet | Part A: Pimasertib Tablet Then Pimasertib Capsule | Part B:Pimasertib Capsule
Started | 0 | 0 | 38
Completed | 0 | 0 | 38
Not Completed | 0 | 0 | 0

BASELINE CHARACTERISTICS:
Population: Safety analysis set included all subjects who received at least one dose of investigational medicinal product (IMP).
Groups:
- Entire Study Population: It included all the subjects randomized to receive either Pimasertib 60 mg capsule and Pimasertib 60 mg tablet first in Part A and Pimasertib 60 mg capsule in Part B of the study.
Arm/Group | Entire Study Population
Number analyzed (Participants) | 38
Age, Continuous [Mean (Standard Deviation); unit: years] | 60.6 (11.74)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 20
  Male | 18

OUTCOME MEASURES:

1. Primary Outcome: Maximum Observed Plasma Concentration (Cmax)
Description: Maximum observed plasma concentration (Cmax) was calculated for Part A Pimasertib 60 mg Capsule and tablet.
Time Frame: Predose, 0.25, 0.5, 0.75, 1, 1.5, 2, 2.5, 4, 8, and 24 hours post-dose on Day 1 and 3
Population: Pharmacokinetic (PK) analysis set included all subjects who received the Part A IMP, had compliance with IMP intake in Part A, at least one post-treatment PK sample from each treatment period and absence of protocol deviations affecting bioavailability.
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: nanogram per milliliter (ng/mL)
Groups:
- Part A: Pimasertib 60 mg Capsule: A single dose of 2 Pimasertib 30 mg capsule administered orally in one of the intervention periods in part A of the study.
- Part A: Pimasertib 60 mg Tablet: A single dose of 3 Pimasertib 20 mg tablet administered orally in one of the intervention periods in part A of the study.
Arm/Group | Part A: Pimasertib 60 mg Capsule | Part A: Pimasertib 60 mg Tablet
Number analyzed (Participants) | 37 | 37
nanogram per milliliter (ng/mL) | 254.6 (75.7) | 314.1 (84.2)

2. Secondary Outcome: Area Under the Plasma Concentration-time Curve From Zero to Infinity (AUC0-inf)
Time Frame: Predose, 0.25, 0.5, 0.75, 1, 1.5, 2, 2.5, 4, 8, and 24 hours post-dose on Day 1 and 3
Population: PK analysis set included all subjects who received the Part A IMP, had compliance with IMP intake in Part A, at least one post-treatment PK sample from each treatment period and absence of protocol deviations affecting bioavailability. Here N (number of participants analysed) signifies the number of subjects analysed for this outcome measure.
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: h*ng/mL
Arm/Group | Part A: Pimasertib 60 mg Capsule | Part A: Pimasertib 60 mg Tablet
Number analyzed (Participants) | 32 | 36
h*ng/mL | 1110.3 (74.2) | 1109.2 (72.9)

3. Secondary Outcome: Time to Reach Maximum Observed Plasma Concentration (Tmax)
Time Frame: Predose, 0.25, 0.5, 0.75, 1, 1.5, 2, 2.5, 4, 8, and 24 hours post-dose on Day 1 and 3
Population: PK analysis set included all subjects who received the Part A IMP, had compliance with IMP intake in Part A, at least one post-treatment PK sample from each treatment period and absence of protocol deviations affecting bioavailability.
Measure: Median (Full Range); unit: hour
Arm/Group | Part A: Pimasertib 60 mg Capsule | Part A: Pimasertib 60 mg Tablet
Number analyzed (Participants) | 37 | 37
hour | 0.750 [0.25 to 4.05] | 0.517 [0.25 to 3.93]

4. Secondary Outcome: Apparent Terminal Half-life (t1/2)
Time Frame: Predose, 0.25, 0.5, 0.75, 1, 1.5, 2, 2.5, 4, 8, and 24 hours post-dose on Day 1 and 3
Population: PK analysis set included all subjects who received the Part A IMP, had compliance with IMP intake in Part A, at least one post-treatment PK sample from each treatment period and absence of protocol deviations affecting bioavailability. Here N (number of participants analyzed) signifies the number of subjects analysed for this outcome measure.
Measure: Median (Full Range); unit: hour
Arm/Group | Part A: Pimasertib 60 mg Capsule | Part A: Pimasertib 60 mg Tablet
Number analyzed (Participants) | 32 | 36
hour | 4.38 [1.65 to 8.15] | 4.47 [0.71 to 6.21]

5. Secondary Outcome: Apparent Total Body Clearance (CL/f)
Description: Clearance of a drug was a measure of the rate at which a drug is metabolized or eliminated by normal biological processes. Drug clearance is a quantitative measure of the rate at which a drug substance is removed from the blood.
Time Frame: Predose, 0.25, 0.5, 0.75, 1, 1.5, 2, 2.5, 4, 8, and 24 hours post-dose on Day 1 and 3
Population: as for outcome 4
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: liter per hour (L/h)
Arm/Group | Part A: Pimasertib 60 mg Capsule | Part A: Pimasertib 60 mg Tablet
Number analyzed (Participants) | 32 | 36
liter per hour (L/h) | 54.041 (74.2) | 54.092 (72.9)

6. Secondary Outcome: Apparent Volume of Distribution (Vz/f)
Description: Volume of distribution was defined as the theoretical volume in which the total amount of drug would need to be uniformly distributed to produce the desired plasma concentration of a drug. Apparent volume of distribution after oral dose (Vz/F) is influenced by the fraction absorbed.
Time Frame: Predose, 0.25, 0.5, 0.75, 1, 1.5, 2, 2.5, 4, 8, and 24 hours post-dose on Day 1 and 3
Population: as for outcome 4
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: Liter
Arm/Group | Part A: Pimasertib 60 mg Capsule | Part A: Pimasertib 60 mg Tablet
Number analyzed (Participants) | 32 | 36
Liter | 346.454 (54.1) | 334.540 (59.0)

7. Secondary Outcome: Terminal Rate Constant (λz)
Time Frame: Predose, 0.25, 0.5, 0.75, 1, 1.5, 2, 2.5, 4, 8, and 24 hours post-dose on Day 1 and 3
Population: as for outcome 4
Measure: Median (Full Range); unit: 1/h
Arm/Group | Part A: Pimasertib 60 mg Capsule | Part A: Pimasertib 60 mg Tablet
Number analyzed (Participants) | 32 | 36
1/h | 0.16 [0.09 to 0.42] | 0.15 [0.11 to 0.98]

8. Primary Outcome: Area Under the Plasma Concentration-time Curve From Zero to the Last Quantifiable Concentration (AUC 0-t)
Description: Area under the plasma concentration-time curve from time zero to the last sampling time (AUC0-t) at which the concentration was at or above the lower limit of quantification.
Time Frame: Predose, 0.25, 0.5, 0.75, 1, 1.5, 2, 2.5, 4, 8, and 24 hours post-dose on Day 1 and 3
Population: as for outcome 3
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: hour*nanogram per milliliter (h*ng/mL)
Arm/Group | Part A: Pimasertib 60 mg Capsule | Part A: Pimasertib 60 mg Tablet
Number analyzed (Participants) | 37 | 37
hour*nanogram per milliliter (h*ng/mL) | 979.0 (76.5) | 1060.7 (73.0)

9. Secondary Outcome: Number of Subjects With Treatment Emergent Adverse Events (TEAEs), Serious TEAEs, and TEAEs Leading to Discontinuation
Description: An AE was any untoward medical occurrence in a subject who received study drug without regard to possibility of causal relationship. An SAE was an AE resulting in any of the following outcomes or deemed significant for any other reason: death; initial or prolonged inpatient hospitalization; life-threatening experience (immediate risk of dying); persistent or significant disability/incapacity; congenital anomaly. Treatment-emergent are events between first dose of study drug administration until 30 days after the last dose of study drug administration that were absent before treatment or that worsened relative to pre treatment state.
Time Frame: From the first dose of study drug administration until 30 days after the last dose of study drug administration, assessed up to 14 Months
Population: Safety analysis set included all subjects who received at least one dose of IMP.
Measure: Number; unit: subjects
Groups:
- Part B: Pimasertib Capsule: Pimasertib 2 capsule 30 mg orally twice daily up to 4 cycles of 21 days each in Part B and trial extension phase until disease progression, intolerable toxicity, subject withdrawal, loss to follow-up or death.
Arm/Group | Part A: Pimasertib 60 mg Capsule | Part A: Pimasertib 60 mg Tablet | Part B: Pimasertib Capsule
Number analyzed (Participants) | 38 | 37 | 38
subjects
  TEAEs | 19 | 20 | 38
  Serious TEAEs | 1 | 0 | 19
  TEAEs leading to discontinuation | 0 | 0 | 13

10. Secondary Outcome: Part B: Number of Subjects Who Experienced Complete Response (CR)
Description: CR as per Response Evaluation Criteria In Solid Tumors (RECIST) v1.1 defined as disappearance of all target lesions except lymph nodes (LN); LN must have a decrease in the short axis to less than (<)10 millimeter (mm).
Time Frame: Screening to Day 1 of each cycle (21 day in each cycle) until disease progression, intolerable toxicity, withdrawal of consent or death; assessed up to 14 Months
Population: Safety analysis set included all subjects who received at least one dose of IMP.
Measure: Number; unit: subjects
Arm/Group | Part B: Pimasertib Capsule
Number analyzed (Participants) | 38
subjects | 0

11. Secondary Outcome: Part B: Number of Subjects Who Experienced Partial Response (PR)
Description: PR as per RECIST v1.1 defined as 30% decrease in sum of diameters of target lesions taking as reference the baseline sum diameters.
Time Frame: as for outcome 10
Population: Safety analysis set included all subjects who received at least one dose of IMP.
Measure: Number; unit: subjects
Arm/Group | Part B: Pimasertib Capsule
Number analyzed (Participants) | 38
subjects | 1

12. Secondary Outcome: Part B: Number of Subjects Who Experienced Stable Disease (SD)
Description: SD as per RECIST v1.1 defined as neither shrinkage to qualify for PR nor increase to qualify for progressive disease (PD) taking the smallest sum diameters on study as reference. PR = 30% decrease in sum of diameters of target lesions taking as reference the baseline sum diameters; PD = 20% increase in sum of diameters of target lesions; the appearance of >=1 new lesions.
Time Frame: as for outcome 10
Population: Safety analysis set included all subjects who received at least one dose of IMP.
Measure: Number; unit: subjects
Arm/Group | Part B: Pimasertib Capsule
Number analyzed (Participants) | 38
subjects | 10

13. Secondary Outcome: Part B: Number of Subjects Who Experienced Progressive Disease (PD)
Description: PD as per RECIST v1.1 defined as 20% increase in sum of diameters of target lesions; the appearance of >=1 new lesions.
Time Frame: as for outcome 10
Population: Safety analysis set included all subjects who received at least one dose of IMP.
Measure: Number; unit: subjects
Arm/Group | Part B: Pimasertib Capsule
Number analyzed (Participants) | 38
subjects | 15

ADVERSE EVENTS:
Time Frame: Baseline up to end of trial (before the start of a new anticancer therapy or 30 ± 2 days after the last investigational medicinal product administration.)
Groups:
- Part B: Pimasertib Capsule (BID): Pimasertib 2 capsule 30 mg orally twice daily up to 4 cycles of 21 days each in Part B and trial extension phase until disease progression, intolerable toxicity, subject withdrawal, loss to follow-up or death.
Arm/Group | Part A: Pimasertib 60 mg Capsule | Part A: Pimasertib 60 mg Tablet | Part B: Pimasertib Capsule (BID)
Serious Adverse Events (participants affected / at risk) | 1/38 | 0/37 | 19/38
Other Adverse Events (participants affected / at risk) | 18/38 | 17/37 | 37/38
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Part A: Pimasertib 60 mg Capsule (N=38) | Part A: Pimasertib 60 mg Tablet (N=37) | Part B: Pimasertib Capsule (BID) (N=38)
Cardiac failure congestive (Cardiac disorders) | 0 | 0 | 1
Diarrhoea (Gastrointestinal disorders) | 1 | 0 | 2
Abdominal pain upper (Gastrointestinal disorders) | 0 | 0 | 1
Gastrointestinal haemorrhage (Gastrointestinal disorders) | 0 | 0 | 1
Rectal haemorrhage (Gastrointestinal disorders) | 0 | 0 | 1
Small intestinal obstruction (Gastrointestinal disorders) | 0 | 0 | 1
Pyrexia (General disorders) | 1 | 0 | 2
Disease progression (General disorders) | 0 | 0 | 1
Fatigue (General disorders) | 0 | 0 | 1
Non-cardiac chest pain (Gastrointestinal disorders) | 0 | 0 | 1
Oedema peripheral (General disorders) | 0 | 0 | 1
Bile duct obstruction (Hepatobiliary disorders) | 0 | 0 | 1
Pneumonia klebsiella (Infections and infestations) | 1 | 0 | 1
Septic shock (Infections and infestations) | 1 | 0 | 1
Bronchitis (Infections and infestations) | 0 | 0 | 1
Pyelonephritis (Infections and infestations) | 0 | 0 | 1
Blood creatine phosphokinase increased (Investigations) | 0 | 0 | 1
Dehydration (Metabolism and nutrition disorders) | 0 | 0 | 1
Malignant ascites (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 0 | 1
Tumour pain (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 0 | 1
Seizure (Nervous system disorders) | 0 | 0 | 1
Syncope (Nervous system disorders) | 0 | 0 | 1
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 1
Hypoxia (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 1
Pleural effusion (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 1
Pneumonitis (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 1
Pneumothorax (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 1
Pulmonary embolism (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 1
Pulmonary hypertension (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 1
Rash (Skin and subcutaneous tissue disorders) | 0 | 0 | 1
Hypertension (Vascular disorders) | 0 | 0 | 2
Hypotension (Vascular disorders) | 0 | 0 | 2
Deep vein thrombosis (Vascular disorders) | 0 | 0 | 1
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Part A: Pimasertib 60 mg Capsule (N=38) | Part A: Pimasertib 60 mg Tablet (N=37) | Part B: Pimasertib Capsule (BID) (N=38)
Iron deficiency anaemia (Blood and lymphatic system disorders) | 1 | 0 | 4
Anaemia (Blood and lymphatic system disorders) | 1 | 0 | 3
Thrombocytopenia (Blood and lymphatic system disorders) | 0 | 0 | 3
Vision blurred (Eye disorders) | 1 | 4 | 7
Retinal detachment (Eye disorders) | 0 | 0 | 9
Visual impairment (Eye disorders) | 2 | 1 | 3
Chorioretinopathy (Eye disorders) | 0 | 0 | 4
Macular detachment (Eye disorders) | 0 | 0 | 4
Dry eye (Eye disorders) | 0 | 0 | 3
Colour blindness acquired (Eye disorders) | 0 | 0 | 2
Periorbital oedema (Eye disorders) | 0 | 0 | 2
Retinal exudates (Eye disorders) | 0 | 0 | 2
Diarrhoea (Gastrointestinal disorders) | 2 | 6 | 22
Nausea (Gastrointestinal disorders) | 3 | 2 | 13
Vomiting (Gastrointestinal disorders) | 1 | 0 | 9
Stomatitis (Gastrointestinal disorders) | 1 | 0 | 7
Constipation (Gastrointestinal disorders) | 0 | 1 | 2
Dry mouth (Gastrointestinal disorders) | 1 | 0 | 2
Abdominal pain (Gastrointestinal disorders) | 0 | 0 | 2
Ascites (Gastrointestinal disorders) | 0 | 0 | 2
Fatigue (General disorders) | 2 | 0 | 20
Oedema peripheral (General disorders) | 0 | 0 | 10
Pyrexia (General disorders) | 1 | 0 | 8
Chills (General disorders) | 1 | 0 | 3
Non-cardiac chest pain (General disorders) | 0 | 0 | 3
Early satiety (General disorders) | 0 | 0 | 2
Urinary tract infection (Infections and infestations) | 0 | 0 | 3
Oral candidiasis (Infections and infestations) | 0 | 0 | 2
Rash pustular (Infections and infestations) | 0 | 0 | 2
Upper respiratory tract infection (Infections and infestations) | 0 | 0 | 2
Blood creatine phosphokinase increased (Investigations) | 0 | 0 | 17
Blood creatinine increased (Investigations) | 1 | 0 | 2
Gamma-glutamyltransferase increased (Investigations) | 0 | 0 | 2
Transaminases increased (Investigations) | 0 | 0 | 2
Decreased appetite (Metabolism and nutrition disorders) | 1 | 0 | 4
Hypomagnesaemia (Metabolism and nutrition disorders) | 0 | 1 | 2
Dehydration (Metabolism and nutrition disorders) | 0 | 0 | 2
Hypokalaemia (Metabolism and nutrition disorders) | 0 | 0 | 2
Hyponatraemia (Metabolism and nutrition disorders) | 0 | 0 | 2
Hypovolaemia (Metabolism and nutrition disorders) | 0 | 0 | 2
Muscular weakness (Musculoskeletal and connective tissue disorders) | 0 | 0 | 4
Arthralgia (Musculoskeletal and connective tissue disorders) | 0 | 0 | 2
Back pain (Musculoskeletal and connective tissue disorders) | 0 | 0 | 2
Dizziness (Nervous system disorders) | 0 | 1 | 7
Headache (Nervous system disorders) | 1 | 0 | 3
Neuropathy peripheral (Nervous system disorders) | 0 | 0 | 3
Syncope (Nervous system disorders) | 0 | 0 | 2
Mental status changes (Psychiatric disorders) | 0 | 0 | 3
Confusional state (Psychiatric disorders) | 0 | 0 | 2
Dyspnoea exertional (Respiratory, thoracic and mediastinal disorders) | 0 | 1 | 6
Cough (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 4
Pleural effusion (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 4
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 1 | 0 | 2
Oropharyngeal pain (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 2
Rash (Skin and subcutaneous tissue disorders) | 1 | 1 | 13
Dermatitis acneiform (Skin and subcutaneous tissue disorders) | 0 | 0 | 6
Rash maculo-papular (Skin and subcutaneous tissue disorders) | 0 | 0 | 5
Pruritus (Skin and subcutaneous tissue disorders) | 0 | 0 | 3
Palmar-plantar erythrodysaesthesia syndrome (Skin and subcutaneous tissue disorders) | 0 | 0 | 2
Rash erythematous (Skin and subcutaneous tissue disorders) | 0 | 0 | 2
Swelling face (Skin and subcutaneous tissue disorders) | 0 | 0 | 2
Hypotension (Vascular disorders) | 2 | 0 | 3
Hypertension (Vascular disorders) | 0 | 0 | 2

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other